CLINICAL TRIAL: NCT01970696
Title: International Ovarian & Testicular Stromal Tumor Registry
Acronym: OTST
Status: Recruiting | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Children's National Research Institute (Other); Dana-Farber Cancer Institute (Other); Washington University School of Medicine (Other); University of Texas Southwestern Medical Center (Other); M.D. Anderson Cancer Center (Other); Children's Hospital Colorado (Other); Rutgers University (Other); Massachusetts General Hospital (Other); Klinikum Dortmund Wirbelsäulenchirurgie (Other); ResourcePath, LLC (Unknown); Allina Health System (Other); Phoenix Children's Hospital (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Kris Ann Schultz, Kris Ann P. Schultz, MD, MS, Children's Hospitals and Clinics of Minnesota
Other Study IDs: International OTST Registry
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Sex-cord Stromal Tumor; Testicular Stromal Tumors; Ovarian Small Cell Carcinoma
Keywords: ovarian; testicular; stromal; sertoli; leydig; juvenile granulosa cell tumor; gynandroblastoma
MeSH Terms: conditions — Sex Cord-Gonadal Stromal Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — 1) whole blood for DNA extraction and lymphoblastoid cell line generation, 2) stained and unstained slides 3) paraffine blocks and/or scrolls 4) snap frozen tumor tissue (if available), and 5) fresh tissue (if available).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ovarian Stromal Tumors
- Testicular Stromal Tumors
- Ovarian Small Cell Carcinoma

SUMMARY:
Rare tumors are understudied, yet have the potential to shed light on vast areas of cancer research. Ovarian sex cord-stromal tumors, rare tumors of childhood and young adulthood, have recently been found to be associated with a lung cancer of early childhood called pleuropulmonary blastoma (PPB). The cause of these ovarian tumors is unknown. DICER1 mutations are seen in the majority of children with PPB. Research shows DICER1 mutations are also seen in some patients with ovarian tumors. Like PPB, ovarian stromal tumors are highly curable when found in early stage; however, later forms of the disease are aggressive and often fatal. The International Ovarian Stromal Tumor Registry collects clinical and biologic data to understand why these tumors occur and how to treat them. Current work involves the study of the role of DICER1 and miRNA expression in ovarian stromal tumors. Understanding the clinical history, predisposing factors and DICER1 and miRNA expression in these ovarian tumors of childhood will lead to targeted screening and risk stratification for evidence-based treatment and biologically rational therapies. These efforts will improve the lives of children by increasing survival and reducing late effects.

The specific goals of the International Ovarian and Testicular Stromal Tumor Registry are:

1. to understand risk factors by studying age, pathologic subtype, histopathologic features, tumor invasiveness, degree of differentiation, presence of metastasis
2. to collect information on personal and family history in order to refine the clinical characteristics of patients and families with and without germline DICER1 mutations and other genetic predisposing factors
3. to determine whether there is a pattern of gene expression or DNA alterations that correlate with predisposition to ovarian tumors, biologic behavior and clinical outcome
4. to determine optimal screening regimens
5. to use clinical data obtained through the Registry to refine treatment algorithms
6. to establish a collection of annotated biology specimens (tumor tissue and germline DNA) for future research

DETAILED DESCRIPTION:
The Registry collects and analyzes case-by-case data on ovarian and testicular stromal tumors. Cases are identified:

1. by referrals from clinicians or pathologists
2. by families initiating contact with the Registry
3. by Registry requests to authors of published cases to share further details

The data collected include:

1. clinical and laboratory findings
2. family history
3. imaging studies
4. surgery records
5. pathology records including review and study of pathology materials
6. treatment (surgery, chemotherapy, radiation)
7. recurrences or metastases
8. long-term follow-up

The demographic and clinical data are abstracted into a database secured by password protection. Each record in the database has a unique Registry number.

Enrollment in the OTST Registry is based on local diagnosis, but central pathology review is offered as a part of Registry procedures.

For each patient enrolled, the Registry will request 1) whole blood for DNA extraction and lymphoblastoid cell line generation 2) slides or snap frozen tumor tissue (if available), 3) paraffin blocks and/or scrolls and 4) fresh tissue. In some cases, saliva samples, buccal swabs or urine samples will be obtained for DNA extraction.

Pathology materials are centrally reviewed when available. Any discrepancies in the diagnostic interpretation are discussed with the submitting pathologist or clinician. When the central review pathologist cannot confirm diagnosis of a stromal tumor, the referring physician is notified. The local pathologist retains responsibility for the final pathological diagnosis. It is the responsibility of the referring physician to notify the patient regarding any discrepancy found.

Biologic specimens will be banked and stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Previous or current diagnosis of an ovarian sex cord stromal including but not limited to: Sertoli-Leydig cell tumor, gynandroblastoma (now enrolling these patients on PPB/DICER1 Registry), juvenile granulosa cell tumor, Sertoli cell tumor, sex cord-stromal tumor with annular tubules or undifferentiated stromal tumor
* Previous or current diagnosis of a testicular stromal tumor including but not limited to: juvenile granulosa cell tumor, Sertoli cell tumor, Leydig cell tumor or undifferentiated stromal tumor

Exclusion Criteria:

* Unable to provide informed consent/assent
* Adult Granulosa cell tumor (unless otherwise specified by Medical Director)

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospectively or retrospectively diagnosed patients with ovarian or testicular stromal tumors or ovarian small cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-12-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
DICER1 mutations in ovarian and testicular stromal tumors | 3 years
  We will analyze germline DNA from patients with gonadal stromal tumors to determine the presence of DICER1 mutations. The tumor tissue will also be sequenced. mRNA and miRNA expression will be analyzed on tumor tissue. Results of the above will be correlated with clinical outcome.

SECONDARY OUTCOMES:
Clinical factors associated with outcome in ovarian and testicular stromal tumors | 10 years
  We will analyze the clinical records to determine which factors influence prognosis
Pathologic and Genetic Correlations | 5 years
  We will correlate the pathologic and genetic data with clinical data to describe factors associated with poor prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann P Schultz, MD, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Schultz KA, Schneider DT, Pashankar F, Ross J, Frazier L. Management of ovarian and testicular sex cord-stromal tumors in children and adolescents. J Pediatr Hematol Oncol. 2012 May;34 Suppl 2:S55-63. doi: 10.1097/MPH.0b013e31824e3867. PMID 22525408
- [Background] Schultz KA, Sencer SF, Messinger Y, Neglia JP, Steiner ME. Pediatric ovarian tumors: a review of 67 cases. Pediatr Blood Cancer. 2005 Feb;44(2):167-73. doi: 10.1002/pbc.20233. PMID 15490488
- [Background] Schultz KA, Ness KK, Nagarajan R, Steiner ME. Adnexal masses in infancy and childhood. Clin Obstet Gynecol. 2006 Sep;49(3):464-79. doi: 10.1097/00003081-200609000-00007. PMID 16885654
- [Background] Rio Frio T, Bahubeshi A, Kanellopoulou C, Hamel N, Niedziela M, Sabbaghian N, Pouchet C, Gilbert L, O'Brien PK, Serfas K, Broderick P, Houlston RS, Lesueur F, Bonora E, Muljo S, Schimke RN, Bouron-Dal Soglio D, Arseneau J, Schultz KA, Priest JR, Nguyen VH, Harach HR, Livingston DM, Foulkes WD, Tischkowitz M. DICER1 mutations in familial multinodular goiter with and without ovarian Sertoli-Leydig cell tumors. JAMA. 2011 Jan 5;305(1):68-77. doi: 10.1001/jama.2010.1910. PMID 21205968
- [Background] Schultz KAP, Stewart DR, Kamihara J, Bauer AJ, Merideth MA, Stratton P, Huryn LA, Harris AK, Doros L, Field A, Carr AG, Dehner LP, Messinger Y, Hill DA. DICER1 Tumor Predisposition. 2014 Apr 24 [updated 2020 Apr 30]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK196157/ PMID 24761742
- [Background] Pappo AS, Furman WL, Schultz KA, Ferrari A, Helman L, Krailo MD. Rare Tumors in Children: Progress Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):3047-54. doi: 10.1200/JCO.2014.59.3632. Epub 2015 Aug 24. PMID 26304909
- [Background] Pashankar F, Bisogno G, Ribeiro R, Messinger Y, Schultz KA, Rodriguez-Galindo C. The role of registries and tumor banking in rare pediatric tumors. Curr Pediatr Rep 2015:1-9. Avail online 15 Mar 2015. DOI 10.1007/s40124-015-0077-9.
- [Background] Schultz KAP and Miller R. (2014) Adnexal Masses in Infancy and Childhood. Coomarasamy A, Davuka W, Shafi M, Chan C (eds): Gynecology and Obstetric Surgery: Challenges and Management Options. Wiley-Blackwell. [BOOK.] [In press; avail may 2015].
- [Background] Schultz KAP, Frazier L, Schneider DT. (2014) Ovarian and Testicular Sex Cord Stromal Tumors. Frazier, AL, Amatruda JF (eds): Textbook Pediatric Germ Cell Tumors, Pediatric Oncology 1. Berlin Heidelberg. Springer-Verlag. [BOOK.].
- [Background] Schneider DT, Orbach D, Ben-Ami T, Bien E, Bisogno G, Brecht IB, Cecchetto G, Ferrari A, Godzinski J, Janic D, Lopez Almaraz R, Pourtsidis A, Roganovic J, Schultz KAP, Stachowicz-Stencel T, Fresneau B. Consensus recommendations from the EXPeRT/PARTNER groups for the diagnosis and therapy of sex cord stromal tumors in children and adolescents. Pediatr Blood Cancer. 2021 Jun;68 Suppl 4:e29017. doi: 10.1002/pbc.29017. Epub 2021 Mar 24. PMID 33760357
- [Result] Doros L, Yang J, Dehner L, Rossi CT, Skiver K, Jarzembowski JA, Messinger Y, Schultz KA, Williams G, Andre N, Hill DA. DICER1 mutations in embryonal rhabdomyosarcomas from children with and without familial PPB-tumor predisposition syndrome. Pediatr Blood Cancer. 2012 Sep;59(3):558-60. doi: 10.1002/pbc.24020. Epub 2011 Dec 16. PMID 22180160
- [Result] Schultz KA, Pacheco MC, Yang J, Williams GM, Messinger Y, Hill DA, Dehner LP, Priest JR. Ovarian sex cord-stromal tumors, pleuropulmonary blastoma and DICER1 mutations: a report from the International Pleuropulmonary Blastoma Registry. Gynecol Oncol. 2011 Aug;122(2):246-50. doi: 10.1016/j.ygyno.2011.03.024. Epub 2011 Apr 17. PMID 21501861
- [Result] Schultz KA, Harris A, Williams GM, Baldinger S, Doros L, Valusek P, Frazier AL, Dehner LP, Messinger Y, Hill DA. Judicious DICER1 testing and surveillance imaging facilitates early diagnosis and cure of pleuropulmonary blastoma. Pediatr Blood Cancer. 2014 Sep;61(9):1695-7. doi: 10.1002/pbc.25092. Epub 2014 May 13. PMID 24821309
- [Result] Schultz KA, Harris A, Messinger Y, Sencer S, Baldinger S, Dehner LP, Hill DA. Ovarian tumors related to intronic mutations in DICER1: a report from the international ovarian and testicular stromal tumor registry. Fam Cancer. 2016 Jan;15(1):105-10. doi: 10.1007/s10689-015-9831-y. PMID 26289771
- [Result] Rutter MM, Jha P, Schultz KA, Sheil A, Harris AK, Bauer AJ, Field AL, Geller J, Hill DA. DICER1 Mutations and Differentiated Thyroid Carcinoma: Evidence of a Direct Association. J Clin Endocrinol Metab. 2016 Jan;101(1):1-5. doi: 10.1210/jc.2015-2169. Epub 2015 Nov 10. PMID 26555935
- [Result] Rove KO, Maroni PD, Cost CR, Fairclough DL, Giannarini G, Harris AK, Schultz KA, Cost NG. Pathologic Risk Factors in Pediatric and Adolescent Patients With Clinical Stage I Testicular Stromal Tumors. J Pediatr Hematol Oncol. 2015 Nov;37(8):e441-6. doi: 10.1097/MPH.0000000000000445. PMID 26479987
- [Result] Golmard L, Vasta LM, Duflos V, Corsini C, Dubois d'Enghien C, McMaster ML, Harney LA, Carr AG, Ling A, Dijoud F, Gauthier A, Miettinen M, Cost NG, Gauthier-Villars M, Orbach D, Irtan S, Haouy S, Schultz KA, Stoppa-Lyonnet D, Coupier I, Stewart DR, Sirvent N. Testicular Sertoli cell tumour and potentially testicular Leydig cell tumour are features of DICER1 syndrome. J Med Genet. 2022 Apr;59(4):346-350. doi: 10.1136/jmedgenet-2020-107434. Epub 2021 Mar 29. PMID 33782093
- [Result] Kebudi R, Dural O, Bay SB, Gorgun O, Onder S, Bilgic B, Yilmaz I, Iribas A, Arndt CA, Harris AK, Field A, Schultz KAP, Hill DA. Childhood Rhabdomyosarcoma of the Female Genital Tract: Association with Pathogenic DICER1 Variation, Clinicopathological Features, and Outcomes. J Pediatr Adolesc Gynecol. 2021 Aug;34(4):449-453. doi: 10.1016/j.jpag.2021.01.011. Epub 2021 Jan 20. PMID 33484847
- [Result] Schneider KW, Cost NG, Schultz KAP, Svihovec S, Suttman A. Germline predisposition to genitourinary rhabdomyosarcoma. Transl Androl Urol. 2020 Oct;9(5):2430-2440. doi: 10.21037/tau-20-76. PMID 33209717
- [Result] Vasta LM, McMaster ML, Harney LA, Ling A, Kim J, Harris AK, Carr AG, Damrauer SM, Rader DJ, Kember RL, Kanetsky PA, Nathanson KL, Pyle LC, Greene MH, Schultz KA, Stewart DR; Regeneron Genetics Center (RGC) Research Team. Lack of pathogenic germline DICER1 variants in males with testicular germ-cell tumors. Cancer Genet. 2020 Oct;248-249:49-56. doi: 10.1016/j.cancergen.2020.10.002. Epub 2020 Oct 24. PMID 33158809
- [Result] Dural O, Kebudi R, Yavuz E, Yilmaz I, Buyukkapu Bay S, Schultz KAP, Hill DA. DICER1-Related Embryonal Rhabdomyosarcoma of the Uterine Corpus in a Prepubertal Girl. J Pediatr Adolesc Gynecol. 2020 Apr;33(2):173-176. doi: 10.1016/j.jpag.2019.12.002. Epub 2019 Dec 12. PMID 31838154
- [Result] Schultz KAP, Harris AK, Finch M, Dehner LP, Brown JB, Gershenson DM, Young RH, Field A, Yu W, Turner J, Cost NG, Schneider DT, Stewart DR, Frazier AL, Messinger Y, Hill DA. DICER1-related Sertoli-Leydig cell tumor and gynandroblastoma: Clinical and genetic findings from the International Ovarian and Testicular Stromal Tumor Registry. Gynecol Oncol. 2017 Dec;147(3):521-527. doi: 10.1016/j.ygyno.2017.09.034. Epub 2017 Oct 14. PMID 29037807
- [Result] Merideth MA, Harney LA, Vyas N, Bachi A, Carr AG, Hill DA, Dehner LP, Schultz KAP, Stewart DR, Stratton P. Gynecologic and reproductive health in patients with pathogenic germline variants in DICER1. Gynecol Oncol. 2020 Mar;156(3):647-653. doi: 10.1016/j.ygyno.2019.12.037. Epub 2020 Jan 15. PMID 31952842
- [Result] Schultz KA, Harris AK, Schneider DT, Young RH, Brown J, Gershenson DM, Dehner LP, Hill DA, Messinger YH, Frazier AL. Ovarian Sex Cord-Stromal Tumors. J Oncol Pract. 2016 Oct;12(10):940-946. doi: 10.1200/JOP.2016.016261. PMID 27858560
- [Result] Rove KO, Maroni PD, Cost CR, Fairclough DL, Giannarini G, Harris AK, Schultz KA, Cost NG. Pathologic Risk Factors for Metastatic Disease in Postpubertal Patients With Clinical Stage I Testicular Stromal Tumors. Urology. 2016 Nov;97:138-144. doi: 10.1016/j.urology.2016.06.066. Epub 2016 Aug 15. PMID 27538802
- [Result] Terry W, Carlisle EM, Mallinger P, Nelson AT, Gordon D, Messinger YH, Field A, Dehner LP, Hill DA, Schultz KAP. Thoracic Sertoli-Leydig cell tumor: An alternative type of pleuropulmonary blastoma associated with DICER1 variation. Pediatr Blood Cancer. 2021 Nov;68(11):e29284. doi: 10.1002/pbc.29284. Epub 2021 Aug 16. PMID 34398502
- [Result] Nelson AT, Harris AK, Watson D, Kamihara J, Chen KS, Stall JN, Devins KM, Young RH, Olson DR, Mallinger PHR, Mitchell SG, Hoffman LM, Halliday G, Suleymanova AM, Glade Bender JL, Messinger YH, Herzog CE, Field AL, Frazier AL, Stewart DR, Dehner LP, Hill DA, Billmire DF, Schneider DT, Schultz KAP. Outcomes in ovarian Sertoli-Leydig cell tumor: A report from the International Pleuropulmonary Blastoma/DICER1 and Ovarian and Testicular Stromal Tumor Registries. Gynecol Oncol. 2024 Jul;186:117-125. doi: 10.1016/j.ygyno.2024.04.005. Epub 2024 Apr 23. PMID 38657450
- See also: International OTST Registry official website — http://www.OTSTregistry.org
- See also: International PPB/DICER1 Registry — http://www.PPBregistry.org